CLINICAL TRIAL: NCT01046292
Title: Effect of Ginkgo Biloba Special Extract LI 1370 on Dual-tasking in Patients With MCI: a Randomized, Double-blind, Placebo-controlled Exploratory Study
Brief Title: Effect of Ginkgo Biloba Special Extract LI 1370 on Dual-tasking in Patients With MCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBE LI 1370
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Gait, Ginkgo biloba, mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginkgo biloba (Experimental)
  Interventions: Drug: Ginkgo biloba
- Placebo control (Placebo Comparator)
  Interventions: Drug: Ginkgo biloba

INTERVENTIONS:
Drug: Ginkgo biloba — The participants will be randomly allocated to either the intervention group or the placebo control group at a ratio of 1:1. After six months, GBE will be administered to all participants for another 6 months for free. The daily administered dose (taken with meals in the morning and evening) will consist of either twice-daily 1 capsule of Symfona® forte 120mg GBE or identically appearing placebo.
  Other Names: Symfona® forte

SUMMARY:
The aim of this study is to evaluate the effects of Ginkgo Biloba Extract (GBE) in executive function-impaired Mild Cognitive Impairment (MCI) patients by assessing gait while walking alone as well as under differing dual-task conditions.

The primary endpoint in the evaluation of GBE efficacy is gait speed. The secondary endpoint is cycle time variability under dual-task conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-85 years
* Swiss German or German speaker
* Completed elementary school
* Impaired executive function (gait speed reduction ≥ 10% under dual-task as compared to normal walking)
* No dementia according to International Classifications of Diseases (ICD)-10 and Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV.
* Cognitive decline (self/informant report or objective task)
* Preserved basic activities of daily living and minimal impairment in complex instrumental functions
* Written informed consent and nihil obstat

Exclusion Criteria:

* Current drug treatment with Warfarin-like drugs (Coumarins or Clopidogrel), however, acetylsalicylic acid 100mg and 300mg is permitted
* Current intake of GBE or during the last 6 months
* Known hypersensitivity to GBE or its constituents
* Regular intake of antipsychotic, anxiolytic or sedative drugs(allowed if clinically stable for at least the past 3 months while under treatment)
* Concomitant gait-relevant disorders: severe cardio/pulmonary/cerebron -vascular disorders, bleeding diathesis, polyneuropathy and severe orthopedic disorders, organic cerebral disease epilepsy, low vision
* Severe medical conditions (e.g. chronic renal insufficiency, severe hepatic disorders,cardio-vascular disease, uncontrolled hypertension, peptic ulcer, malignoma)
* Participation in another clinical intervention study within the last 2 months
* Use of walking aid
* Normal walking speed is < 100cm/s

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
gait speed | baseline, 3, 6, 12 months

SECONDARY OUTCOMES:
cycle time variability | baseline, 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Reto W Kressig, MD, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Basel University Hospital, Basel Mobility Center, Basel, Canton of Basel-City, Switzerland